CLINICAL TRIAL: NCT05406362
Title: A Randomised, Placebo Controlled, Double Blind, Multicentre Proof of Concept Study to Assess the Safety and Efficacy of Two Doses of VAD044 in Patients With Hereditary Hemorrhagic Telangiectasia (HHT)
Brief Title: Assess Safety and Efficacy of VAD044 in HHT Patients
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Vaderis Therapeutics AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VAD044C002
Record Dates: First submitted 2022-05-10; First posted 2022-06-06 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-02

CONDITIONS: Hereditary Hemorrhagic Telangiectasia (HHT)
Keywords: Osler-Weber-Rendu disease; Arteriovenous Malformations
MeSH Terms: conditions — Telangiectasia, Hereditary Hemorrhagic; Arteriovenous Malformations

STUDY DESIGN:
Intervention Model Description: The patients will be randomised into VAD044 30 mg or 40 mg or placebo group in the ratio 1:1:1, according to a centralised randomisation process
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 30 mg (Experimental): 30 mg VAD044
  Interventions: Drug: VAD044 Part I; Drug: VAD044 Part II
- 40 mg (Experimental): 40 mg VAD044
  Interventions: Drug: VAD044 Part I; Drug: VAD044 Part II
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: VAD044 Part I

INTERVENTIONS:
Drug: VAD044 Part I — capsules to be taken once daily for 12 weeks
  Other Names: VAD044 L-Tartrate gelatin capsules
Drug: VAD044 Part II — capsules to be taken once daily for 12 months
  Other Names: VAD044 L-Tartrate gelatin capsules
  Arms: 30 mg; 40 mg

SUMMARY:
Part I: The purpose of this Phase 1b proof of concept study, randomised, placebo controlled, double blind, multicentre study is to asssess safety and efficacy of 2 doses of VAD044 in adult HHT patients.

Part II: The purpose of this open-label extension following the completion of the randomised double blind treatment and follow-up period (Part I of the study) is to assess the long-term safetty, tolerability and efficacy of VAD044 in adult HHT patients.

DETAILED DESCRIPTION:
Part I: After being informed about the study and the potential risks, all patients giving written informed consent will undergo a two months screening and observation period to determine eligibility for study entry. At Day 0, patients who meet the eligibility requirements will be randomized in a double-blind manner (participant and investigator) in a 1:1:1 ratio to 30mg VAD044 (once daily), 40 mg (once daily) or placebo (once daily).

Part II: Patients who have completed the study Part I can participate in the open-label extension study (Part II).The patients can roll over immediately after last visit of the Part I or at any time at their convenience and according to their availability, but within a timeframe no longer than 8 months after the last visit (visit 12) of the part I. All patients in Part II will receive 30 mg of VAD044 once daily for the first 4 weeks afterwards the daily dose can be increased to 40 mg daily for up to 12 months.

ELIGIBILITY:
For Part I of the study:

Inclusion Criteria:

* Diagnosis of HHT by the Curaçao criteria
* Several epistaxis/week
* Anaemia
* COVID-19 vaccination or positive COVID-19 antibody test
* Patient has given written informed consent to participate in Part I

Exclusion Criteria:

* Type 1 diabetes or uncontrolled type II diabetes (insulin or non-insulin dependent)
* Active COVID-19 infection
* active uncontrolled infection or known to be serologically positive for HIV, Hep B, Hep C infection
* Recent procedures on nasal telangiectases (<6 weeks)
* Requiring therapeutic anticoagulation
* Use of drugs with anti-angiogenic properties in the past 8 weeks
* laboratory abnormalities

Fort Part II of the study:

Inclusion Criteria:

* Completion of Part I of the study
* All adverse events or serious adverse events occuring during Part I of the study have resolved
* Patient has given written informed consent to participate in Part II

Exclusion Criteria:

- Same as in Part I.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-07-18 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Part I: Safety and Tolerability | 12 weeks
  Type and severity of Adverse Events (AEs)
Part II: Safety and Tolerability | 12 months
  Type and severity of Adverse Events (AEs)

SECONDARY OUTCOMES:
Part I: Change in Epistaxis episodes | 12 weeks
  The number of Epistaxis episodes
Part I: Change in Epistaxis duration | 12 weeks
  Epistaxis duration
Part I: Change in Epistaxis intensity | 12 weeks
  Epistaxis flow intensity
Part I: Change in Epistaxis Severity Score (ESS) | 12 weeks
  ESS used to evaluate the current severity of HHT patient nosebleeds (typically in the last three months) and can help health care providers to evaluate how a patient is responding to treatment. This score ranges from 0-10 and is automatically calculated after answering six simple questions. The higher the score the more severe.
Part I: Change in Haemoglobin | 12 weeks
  Haemoglobin
Part I: Change Ferritin | 12 weeks
  Ferritin
Part I: Change in blood Transferrin saturation level | 12 weeks
  Transferrin saturation level
Part I: Change in Iron supplementation needs | 12 weeks
  Iron supplementation needs
Part I: Change Blood tranfusions requirements | 12 weeks
  Blood tranfusions requirements
Part I: Change in the Nasal Outcome for Epistaxis in Hereditary Hemorrhagic Telangiectasia score | 12 weeks
  The Nasal Outcome for Epistaxis in Hereditary Hemorrhagic Telangiectasia (NOSE HHT questionnaire) wil be used to measure physical, social and emotional impacts of epistaxis. It is a 29-items questionnaire using a Likert scale. A higher score indicates a worse outcome
Part I: Quality of Life Scale SF-12 | 12 weeks
  The SF-12 Quality of Life Scale is a scale to evaluate quality of life using 12 questions. In the SF-12, physical (SF12-PCS) and mental (SF12-MCS) component summary scores are calculated as sub-dimensions. The total score of the physical and mental component summary of the scale varies between 0-100. An increase in the score indicates well-being, and a decrease indicates a state of disability.
Part I: Plasma concentration of VAD044 | 12 weeks
  Plasma concentration of VAD044
Part I: Maximum concentration (Cmax) of VAD04 | 12 weeks
  Maximum concentration (Cmax) of VAD044
Part I: Time of maximum concentration (Tmax) of VAD044 | 12 weeks
  Time of maximum concentration (Tmax) of VAD044
Part I: Area under the curve (exposure to drug) during 24 hours (AUC0-24h) of VAD044 | 12 weeks
  Area under the curve (exposure to drug) during 24 hours (AUC0-24h) of VAD044
Part I: Trough concentration (Ctrough) of VAD044 | 12 weeks
  Trough concentration (Ctrough) of VAD044
Part I: Pharmacodynamics (PD) of VAD044 | 12 weeks
  PRP assay to measure the levels of pAKT in the blood in a subset of patients
Part II: Change in The number of Epistaxis episodes | 12 months
  The number of Epistaxis episodes
Part II: Change in Epistaxis duration | 12 months
  Epistaxis duration
Part II: Change in Epistaxis flow intensity | 12 months
  Epistaxis flow intensity
Part II: Change in Epistaxis Severity Score (ESS) | 12 months
  ESS used to evaluate the current severity of HHT patient nosebleeds (typically in the last three months) and can help health care providers to evaluate how a patient is responding to treatment. This score ranges from 0-10 and is automatically calculated after answering six simple questions. The higher the score the more severe.
Part II: Change in Haemoglobin | 12 months
  Haemoglobin
Part II: Change in Ferritin | 12 months
  Ferritin
Part II: Change in Transferrin saturation level | 12 months
  Transferrin saturation level
Part II: Change in Iron supplementation needs | 12 months
  Iron supplementation needs
Part II: Change in blood tranfusions requirements | 12 months
  blood tranfusions requirements
Part II: Quality of Life Scale SF-12 | 12 months
  The SF-12 Quality of Life Scale is a scale to evaluate quality of life using 12 questions. In the SF-12, physical (SF12-PCS) and mental (SF12-MCS) component summary scores are calculated as sub-dimensions. The total score of the physical and mental component summary of the scale varies between 0-100. An increase in the score indicates well-being, and a decrease indicates a state of disability.

CONTACTS AND LOCATIONS:
Overall Officials: Damien Picard, Study Director — Vaderis Therapeutics AG
Locations (7):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- Universitair Ziekenhuis Gent, Ghent, Belgium
- Hospices Civils de Lyon, Lyon, France
- Ospedale Maggiore di Crema, Crema, Italy
- St. Antonius Hospital, Nieuwegein, Netherlands
- Spain (2):
  - Hospital Universiati De Bellvitge, Barcelona
  - Hospital Universitario Ramón y Cajal, Madrid

REFERENCES:
- [Derived] Al-Samkari H, Hessels J, Riera-Mestre A, Dupuis-Girod S, Van Zele T, Gomez Del Olmo V, Hodges PG, Torres-Iglesias R, Berte R, Saint-Mezard P, Lazar H, Benedict N, Barker D, Bernasconi C, Picard D, Buscarini E, Mager HJ. Engasertib versus Placebo for Bleeding in Hereditary Hemorrhagic Telangiectasia. N Engl J Med. 2025 Nov 27;393(21):2131-2141. doi: 10.1056/NEJMoa2504411. PMID 41297007